CLINICAL TRIAL: NCT03791983
Title: Precision Medical Diagnosis and Acupuncture Treatment for Parkinson's Disease -The Evaluation of Scalp Acupuncture for Parkinson's Disease
Brief Title: Precision Medical Diagnosis and Acupuncture Treatment for Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-10-002B
Record Dates: First submitted 2019-01-01; First posted 2019-01-03 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy Group (Experimental)
  Interventions: Other: Scalp Acupuncture
- Control Group (Other)
  Interventions: Other: Body Acupenture

INTERVENTIONS:
Other: Scalp Acupuncture — Scalp acupuncture is a form of alternative medicine in which thin needles are inserted into the scalp. It is a key component of traditional Chinese medicine (TCM).
  Arms: Therapy Group
Other: Body Acupenture — Acupuncture is a form of alternative medicine in which thin needles are inserted into the body. It is a key component of traditional Chinese medicine (TCM).
  Arms: Control Group

SUMMARY:
This study integrates traditional Chinese medicine syndromes and pulse diagnosis, and uses laser vibration overlay and functional cerebral angiography to understand the efficacy of scalp acupuncture against Parkinson's Disease.

DETAILED DESCRIPTION:
Traditional Chinese medicine does not have the term " Parkinson's disease". According to the symptoms of the disease, it is closer to the "Liver wind", "Vibration" and "Chatter" in Chinese medicine. Scalp needle stimulation can increase the content of dopamine in the brain and improve mitochondrial function and reduce the death of substantia nigra.

This study integrates TCM syndromes and pulse diagnosis, and uses laser vibration overlay and functional brain image to understand the effect of scalp acupuncture on Parkinson's disease. The project will be carried out in two phases: the first phase is the pilot study, and 200 patients with limb shakes were collected from the neurology clinic. After the laser vibration overlay test, 20 patients with mild tremors and diagnosed as Parkinson's disease were selected. , treated by Wen's scalp acupuncture. In the second phase, 80 Parkinson patients were enrolled, randomized to the treatment group and the control group, and the changes in TCM syndrome, pulse diagnosis and Parkinson scale were compared before and after treatment, and the fMRI and vibration overlay ratios were evaluated after scalp acupuncture.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as Idiopathic Parkinsonism by Neurologist
2. Have taken first line drugs more than three months
3. Did not take any acupuncture or rehabilitation
4. Voluntary

Exclusion Criteria:

1. Taking anticancer drug now or diagnosed as depression, psychosis or other mental illnesses
2. Medical history of stroke or dementia
3. Taking anticoagulant now or having coagulation disorders
4. Scalp infection
5. Pregnant women
6. Patient with irregular heartbeat, implanted artificial cardiac pacemaker or implanted cardioverter-defibrillator
7. Belonephobia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale | 2 Months
  A comprehensive assessment of both motor and non-motor symptoms associated with Parkinson's. The Unified Parkinson's Disease Rating Scale is made up of 42 items. These items are divided into six sections which are separately "evaluation of mentation, behavior, and mood", "self-evaluation of the activities of daily life", "clinician-scored monitored motor evaluation", "complications of therapy", "Hoehn and Yahr staging of severity of Parkinson's disease" and "Schwab and England ADL scale".The evaluation score for the first item to the 39th item is 0 to 4 points. The evaluation score for the 40th to the 42th item is 0 to 1 points.The higher score meand the worse condition. The sum of all the items'score is the score of the scale. Highr Rating Scales'scores indicate severe symptoms.
Micro Vibration Scan | 2 Months
  1. Discover early symptom before the onset.
  2. Recognize PD tremor pattern within 1 minute.
  3. Non-invasive, Non-radiation, and Low-cost medical device for daily tracking and treatment evaluation.
SPECT | 2 Months
  A type of nuclear imaging test that shows how blood flows to tissues and organs.
PET/MRI | 2 Months
  PET/MRI combines time-of-flight PET with 3-Tesla MRI for exceptional image quality, more conclusive diagnosis, and lower radiation in a single exam. The powerful combination of molecular, functional and anatomic information provides essential data for critical treatment decisions.

SECONDARY OUTCOMES:
Constitution in Chinese Medicine Questionnaire (CCMQ) | 2 Months
  Sixty items were applied to measure the nine constitutions: Neutral (a normal constitution), Qi-deficiency constitution, Yang-deficiency constitution, Yin-deficiency constitution, Phlegm-dampness constitution, Damp-heat constitution, Stagnant-blood constitution, Stagnant-Qi constitution, and Inherited-special constitution.
Sphygmograph | 2 Months
  Diagnoses patient's pulse change

CONTACTS AND LOCATIONS:
Overall Officials: Fang-Pei Chen, MD, Study Chair — Taipei Veterans General Hospital, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided